CLINICAL TRIAL: NCT05024383
Title: Dissecting the Heterogeneity of Oral Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NYU College of Dentistry (Other)
Responsible Party: Principal Investigator, Brian L. Schmidt, Director of Bluestone Center for Clinical Research, NYU College of Dentistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: i21-00964
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Single arm study design with group comparisons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chemical sensitivity — Chemical sensitivity will be evaluated with paper taste strips embedded with varying concentrations of capsaicin solutions (activates TRPV1) and allyl isothiocyanate solutions (activates TRPA1) applied to the tongues of healthy subjects and site of cancer in oral cancer patients.
Other: Mechanical sensitivity — Mechanical sensitivity will be evaluated via von Frey filaments applied to the tongues of healthy subjects and and site of cancer in oral cancer patients.

SUMMARY:
Oral squamous cell carcinoma (SCC) produces a higher prevalence and more severe pain than all other cancers. Orofacial pain is one of the most common initial symptoms of oral cancer and often leads to the diagnosis of oral cancer. However, the character, severity, and unique features of oral cancer widely differ between patients. There is currently no effective and lasting treatment available to alleviate suffering from oral cancer pain.

A significant obstacle to effectively treating cancer pain is that the relative contributions of nociceptive mediators and their mechanisms of action (i.e., responsible receptors) are largely unknown. There is, therefore, a critical need to define the neurobiologic mechanisms responsible for oral cancer pain. Without such information, the promise of non-opioid therapy for the treatment of oral cancer pain will remain unfulfilled.

The primary objective of this study is to define and quantify the phenotype of oral cancer pain in patients, by comparing mechano- and chemosensitivity in oral cancer patients with healthy subjects. Pain will be stimulated on the site of cancer in 40 oral cancer patients and on the tongue in 40 healthy volunteers utilizing chemical sensitivity and mechanical sensitivity tests.

DETAILED DESCRIPTION:
Oral squamous cell carcinoma (SCC) is the sixth most common cancer worldwide. The majority of patients with oral SCC suffer from severe, chronic, function-induced pain. Despite the severity of pain in many patients, the presentation of oral cancer pain is variable. Opioids are the only treatment available for oral cancer pain. Opioids are often ineffective and associated with tolerance, constipation, somnolence, respiratory depression, and addiction, which is now a national crisis.

The current hypothesis for the etiology of oral cancer pain, which is based on clinical studies utilizing questionnaires and preclinical studies, is that cancer cells and cells within the microenvironment produce mediators that activate and sensitize nociceptors. Published and preliminary data indicate that cancer-secreted mediators induce mechano- and chemosensitivity. For example, preliminary clinical studies demonstrate that oral cancer patients experience preoperative sensitivity to capsaicin (i.e., chemosensitivity) and report greater functional (i.e., mechanosensitivity) pain. Capsaicin activates transient receptor potential vanilloid 1 (TRPV1). TRPV1 is activated by temperatures above 43°C and endogenous lipid metabolic products. Mice deficient in TRPV1 respond to mechanical stimuli, suggesting that TRPV1 is not involved in the detection of mechanical stimulation. By contrast, TRP ankyrin repeat 1 (TRPA1), co-localized with TRPV1, is responsive to mechanical stimuli, in addition to irritants such as allyl isothiocyanate (AITC). Both TRPV1 and TRPA1 have been reported to play important roles in orofacial pain. Improved knowledge of the contribution of TRPV1 and TRPA1 to oral cancer pain holds considerable promise for the development of novel, non-opioid treatment strategies that specifically address the unique pain experience of individual patients.

There is a lack of published data characterizing the sensory phenotype of tumor-related cancer pain, which has significant implications for understanding the underlying pathophysiological mechanisms of cancer pain. Quantitative sensory testing can provide insight into the mechanism(s) responsible for pain. In this proposal, we will test our hypothesis that the quality of pain experienced by oral cancer patients is dependent on the level of activation of specific channels on nociceptors. We will perform mechanical (von Frey testing) and chemical sensitivity tests (sensitivity to capsaicin, TRPV1 agonist, and AITC (TRPA1 agonist) on oral cancer patients, and compare the sensitivities to healthy subjects. For cancer patients, we will administer the validated University of California San Francisco (UCSF) Oral Cancer Pain Questionnaire to evaluate the correlation between mechanical and chemical thresholds with relevant aspects of pain.

We propose that the quality of pain experienced by oral cancer patients is quantifiable and dependent on the level of sensitization and activation of specific channels on nociceptors.

ELIGIBILITY:
Inclusion Criteria (oral cancer patients):

* Biopsy-proven squamous cell carcinoma (SCC) of the oral cavity that requires surgical resection
* Lesion is at least 1 cm in greatest surface dimension

Exclusion Criteria (oral cancer patients):

* History of prior surgical, chemotherapeutic, or radiation treatment for head and neck cancer
* Pregnancy or lactation

Inclusion Criteria (healthy subjects):

* In good general health as evidenced by medical history

Exclusion Criteria (healthy subjects):

* Clinically and/or histologically proven oral pre-cancer, oral cancer
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mechanical Sensitivity | Baseline visit
  Pain will be evaluated using verbal feedback from participants for mechanical sensitivity testing.
Chemical Sensitivity | Baseline visit
  Pain will be evaluated using a visual analogue scale for chemical sensitivity testing.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University College of Dentistry, New York, New York, United States

REFERENCES:
- [Background] Schmidt BL, Hamamoto DT, Simone DA, Wilcox GL. Mechanism of cancer pain. Mol Interv. 2010 Jun;10(3):164-78. doi: 10.1124/mi.10.3.7. PMID 20539035
- [Background] Schmidt BL. The neurobiology of cancer pain. Neuroscientist. 2014 Oct;20(5):546-62. doi: 10.1177/1073858414525828. Epub 2014 Mar 24. PMID 24664352
- [Background] Yang F, Zheng J. Understand spiciness: mechanism of TRPV1 channel activation by capsaicin. Protein Cell. 2017 Mar;8(3):169-177. doi: 10.1007/s13238-016-0353-7. Epub 2017 Jan 2. PMID 28044278
- [Background] Jordt SE, Bautista DM, Chuang HH, McKemy DD, Zygmunt PM, Hogestatt ED, Meng ID, Julius D. Mustard oils and cannabinoids excite sensory nerve fibres through the TRP channel ANKTM1. Nature. 2004 Jan 15;427(6971):260-5. doi: 10.1038/nature02282. Epub 2004 Jan 7. PMID 14712238